CLINICAL TRIAL: NCT03687385
Title: The Comparison of Low- and High-flow Nasal Oxygenation to the Blood Oxygen Saturation During Analgo-sedation in ASA Risk Class I, II and III Normal Weight Patients: Randomized Controlled Trial
Brief Title: The Effect of High-flow Nasal Oxygenation to the Saturation During Analgo-sedation in Different ASA Risk Class Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anita Vukovic (Other)
Collaborators: General Hospital Dubrovnik (Other); Clinical Hospital Centre Zagreb (Other)
Responsible Party: Sponsor-Investigator, Anita Vukovic, MD, specialist of anesthesiology, reanimatology and intensive care, University of Split, School of Medicine
Organization: University of Split, School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-285/8-3-17
Record Dates: First submitted 2018-09-21; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Noninvasive Ventilation; Respiratory Insufficiency; Deep Sedation; Hypoxia; Airway Management; Colonoscopy
Keywords: "Noninvasive Ventilation"[Mesh]; "Airway management"[Mesh]; "Adult"[Mesh]; "Colonoscopy"[Mesh]; "Deep Sedation"[Mesh]; "Hypoxia"[Mesh]
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Intervention Model Description: We plan to conduct prospective, parallel group, randomized controlled clinical trial.
  In total, 126 participants will be included in this trial. These participants are patients scheduled for outpatient colonoscopy in analgo-sedation.
  This study includes 126 normal weight patients of anesthesia risk ASA class I, II or III divided in three groups of 42. Each group will be divided in control subgroups of 21 patients who will receive low-flow nasal oxygenation (LFNO) and intervention subgroups of 21 patients who will receive high-flow nasal oxygenation (HFNO) during standardized intravenous analgo-sedation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Anesthesiologist who interviews and examines patients scheduled for colonoscopy under analgo-sedation will enroll eligible participants and will offer procedure explanation and possibility to sign uniformed written consent. Unique personal hospital admission number (UPHAN) will be assigned to all eligible participants. After that, they will be randomized to control or intervention group by using random numbers generator. Anesthesiologist who implements anesthesia will receive nontransparent envelope with assigned intervention provided by independent investigator and will not decide which participant will receive LFNO or HFNO. However, attending anesthesiologist and participants will unavoidably be aware of type of oxygenation applied. Investigator who collects data after procedure will be unaware of study protocol and will enter data to formatted database. Participants' data will be noted under UPHAN. Outcome assessors will be unaware of intervention applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ASA I / LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: low-flow nasal oxygenation (LFNO)
- ASA II / LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: low-flow nasal oxygenation (LFNO)
- ASA III / LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: low-flow nasal oxygenation (LFNO)
- ASA I / HFNO (Experimental): High-flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: high-flow nasal oxygenation (HFNO)
- ASA II/ HFNO (Experimental): High-flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: high-flow nasal oxygenation (HFNO)
- ASA III/ HFNO (Experimental): High-flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: high-flow nasal oxygenation (HFNO)

INTERVENTIONS:
Device: high-flow nasal oxygenation (HFNO) — Experimental HFNO: O2 flow 40L/min, FiO2 40%
  Arms: ASA I / HFNO; ASA II/ HFNO; ASA III/ HFNO
Device: low-flow nasal oxygenation (LFNO) — Active comparator LFNO: O2 flow 5L/min, FiO2 40%
  Arms: ASA I / LFNO; ASA II / LFNO; ASA III / LFNO

SUMMARY:
Analgo-sedation is standard procedure in anesthesiology practice and is often given for colonoscopy in the setting of daily hospital. Ideally, patients should be sedated with preserved spontaneous breathing and adequate blood O2 saturation. To maintain adequate oxygenation, low-flow O2 (2-6 L/min) is usually delivered through standard nasal catheter which can provide inspired fraction (FiO2) of 40% (low-flow nasal oxygenation - LFNO). Coldness and dryness of LFNO applied may be uncomfortable to patient. Standardly applied intravenous anesthetics can lead to transient ceasing of breathing and O2 desaturation despite LFNO. Respiratory instability can also potentiate circulatory instability - undesirable changes in heart rate (HR) and blood pressure (BP). Unlike LFNO, high-flow heated and humidified nasal oxygenation (HFNO) is characterized by the oxygen-air mixture flow of 20 to 70 L/min up to 100% FiO2. Warm and humidified O2, delivered via soft, specially designed nasal cannula, is pleasant to patient. HFNO develops continuous positive pressure of 3 to 7 cmH2O in upper airway which enables noninvasive support to patient's spontaneous breathing thus prolonging time of adequate O2 saturation.

Aim of this study is to compare effect of HFNO and LFNO on oxygenation maintenance before, during and after standardized procedure of intravenous analgo-sedation in normal weight patients of ASA risk I, II and III.

Investigators hypothesize that application of HFNO compared to LFNO, in patients with preserved spontaneous breathing during procedural analgo-sedation, will contribute to maintaining of adequate oxygenation, consequentially adding to greater circulatory and respiratory patients' stability.

Investigators expect that patients who receive HFNO will better maintain adequate oxygenation regarding improved spontaneous breathing. Also patients will have shorter intervals of blood oxygen desaturation, less pronounced rise in blood CO2 level and lesser fall of blood O2 level, less change in HR and BP. Investigators will have to exactly estimate partial and global respiratory insufficiency (blood CO2 and O2 levels) associated with LFNO and HFNO, which will be done by blood-gas analysis of 3 arterial blood samples collected before, during and after analgo - sedation via previously, in local anesthesia, placed arterial cannula. Possible complications will be explained in written uniformed consent and by anesthesiologist.

DETAILED DESCRIPTION:
Analgo-sedation is standard procedure in anesthesiology practice and is often given for diagnostic and procedural intervention in the setting of daily hospital. Institution of sedation and maintaining spontaneous breathing are main characteristics of analgo-sedation. Preservation of adequate patient oxygenation is set up by continuous administration of sedative anesthetic infusion which contributes to hemodynamic stability and by administration of oxygen. Patient oxygenation is implemented prior to analgo-sedation (preoxygenation), during analgo-sedation (periprocedural oxygenation) and during awakening from analgo-sedation (postprocedural oxygenation) usually via nasal cannula with application of low-flow (2-6 L/min) up to 40% of inspired fraction of oxygen (LFNO: low-flow nasal oxygenation, FiO2: inspiratory fraction of oxygen). Despite oxygenation administered, intravenously applied analgo-sedation yields to risk of transitory apnea accompanied by hypoxemia, hypoxia, hypercapnia and hemodynamic insufficiency. Anesthesia risk is classified as ASA classification by American Society of Anesthesiologist Physical Status Classification System: ASA I includes healthy patients without systemic disease, ASA II patients who have mild systemic disease without functional organ limitations and ASA III patients with one or more organ function insufficiency.

High-flow heated and humidified oxygenation (HFNO) delivered via soft, specially designed, nasal cannula is successfully used for preoxygenation of patient with predicted difficulty in ensuring airway patency. Unlike LFNO, HFNO is characterized by high flow of heated and humidified oxygen-air mixture (20-70 L/min) up to 100% FiO2. HFNO prolongs adequate oxygenation time in patients during retrograde endoscopic cholangiopancreatography. Also, HFNO could be alternative for noninvasive ventilation of patients with acute hypoxemic respiratory failure. According to previously mentioned statements, LFNO has significant limitations. Main characteristic of HFNO as innovative technique is supporting patients' spontaneous inspiration effort through high-flow of heated and humidified oxygen-air mixture. Higher inspiratory fraction of oxygen, positive end-expiratory pressure, decreasing of pharyngeal airway dead space and decreasing of airway resistance lead to improved maintaining of oxygenation combined with better patients' tolerance.

AIM of this study is to compare effect of HFNO and LFNO during standardized procedure of intravenous analgo-sedation on periprocedural oxygenation maintenance in normal weight patients of ASA I, II and III status.

Investigators hypothesized that application of HFNO compared to LFNO, in patients with preserved spontaneous breathing during procedural analgo-sedation, contributes to maintaining adequate oxygenation, consequently adding to greater peri-procedural circulatory and respiratory stability of these patients. Investigators expect that HFNO will ensure reduced bradypnoea intervals (frequency of breathing, FoB 1/min), longer maintenance of adequate oxygenation, shorter intervals of desaturation (SpO2 ≤ 92%), reducing hypercapnia (PaCO2 ≥ 6 kPa) and less airway - opening maneuvers performed by attending anesthesiologist (Aom). These will prevent partial respiratory insufficiency detected by low SpO2 or low PaO2 ≤ 11kPa accompanied by normal or low PaCO2 ≤ 6 kPa, and global respiratory insufficiency detected by decreased SpO2 ≤ 92% and PaO2 ≤ 11kPa with increased PaCO2 ≥ 6 kPa.

Investigators plan to conduct prospective, parallel group, randomized controlled clinical trial. Trial will be managed according to principles of Declaration of Helsinki for scientific clinical research and will be planned and guided according to CONSORT guidelines (Consolidated Standards of Reporting Trials). The trial has been approved by hospital's Ethic Committee.

The source of information are going to be 126 adult patients scheduled for colonoscopy under analgo-sedation in the setting of daily outpatient gastroenterology ambulance. Eligible participants will be interviewed and examined ambulatory by anesthesiologist together with evaluation of ASA status, difficulty of airway management and body mass index (BMI). After initial examination inclusive and exclusive criteria will be distinguished. Eligible participants who give their written consent of participation will be included in this study. After that, participants will be assigned to equal ASA I, II or III risk class group. Each group will be randomized to intervention (HFNO) and control (LFNO) subgroup by random numbers generator. Randomization will be used until we reach adequate number of participants in every group.

Interventions: intervention subgroups participants will be oxygenated via nasal cannula using high flow (40 L/min) of humidified and heated oxygen in air mixture (FiO2 40%). HFNO will be applied by oxygenator (AirVO™2, Fisher and Paykell, New Zealand, Technomedika Croatia d.o.o.) during procedural analgo-sedation for colonoscopy with maintained spontaneous breathing. In control subgroups, LFNO will be applied via nasal catheter (Bauerfeind d.o.o, Zagreb, Croatia) using standard low flow oxygen - 5 L/min, FiO2 40%. In both groups concentration of oxygen delivered depends on oxygen flow which is regulated by standard flow-regulator (flowmeter). Oxygen is delivered through pipelines from central hospital gas supply or from portable cylinder gas supply.

Anesthesia procedure will be uniformed for all participants. Integrated noninvasive monitoring of vital functions will be set: EKG - (heart rate/min), SpO2 (%), blood pressure (mmHg), respiratory rate (number of breaths/min) (Compact 7; Medical Econet GmbH, Germany).

Every participant will have established intravenous infusion of 250 ml NaCl 0.9% through intravenous cannula regulated by continuous flow (Extension set/CONTROL-A-FLO Regulator 19" Male Luer Lock Adapter, Baxter/Agmar d.o.o. United States of America/Croatia).

Arterial cannula (REF30401, 20 G - 1,10 mm x 45 mm 49 ml, atraumatic needle tip, Medbar LTD, Izmir, Turkey) will be placed in radial artery in a previously anesthetized area with local anesthetic (EMLA).

Oxygenation (HFNO or LFNO) will be administrated in continuity until patients' awakening. It will be started 3 minutes before starting analgo-sedation (preoxygenation), continued during analgo-sedation and procedure of colonoscopy (perioperative oxygenation) and up to five minutes after colonoscopy and until patient is awake (postprocedural oxygenation).

Intravenous analgo-sedation will be started through continuous infusions of propofol and fentanyl. Induction of sedation will be guided by TCI (Target control Infusion) (B. Braun Melsungen, Germany) with initial target propofol concentration of 6 micrograms/minute. Expected time of induction with this concentration is 60-120 seconds. This target concentration allows hemodynamic and respiratory stability. Required analgesia will be simultaneously applied through slow continuous infusion in dose of 0.05 mcg/kg/min in order to preserve spontaneous breathing. Slow infusion will be applied through perfusor (B.Braun, Melsungen, Germany). Analgo-sedation will be discontinued immediately after end of the procedure.

Control of nasopharyngeal airway passage during procedure is achieved by using oropharyngeal airway, if necessary. Oropharyngeal airway (Airway; Vigon-Medicpro d.o.o.) will be inserted after achieving moderate sedation, and only if base of tongue is closing airway by dropping on posterior pharyngeal wall. Every manipulation of patients' airway by anesthesiologist will be documented (insertion of airway, jaw thrust maneuver).

Sampling: one milliliter of arterial blood will be collected as three consecutive samples from arterial cannula before, during and after analgo-sedation. Sample of arterial blood will be drawn from left radial or cubital artery.

Measurements: measurement of oxygenation will be done using two methods: indirect (noninvasive) method using pulse oxymeter (Compact 7, Medical ECONET GmbH, Germany) and direct (invasive) method from obtained arterial blood sample. Measurement of SpO2 and drawing arterial blood sample will be done simultaneously. Direct measurements of SpO2 and PaO2 will be measured in intervals of time. SpO2 will be measured on the left-hand index finger. Data will be uniformly collected through indirect - noninvasive (SpO2, heart rate, blood pressure, respiratory rate) and direct - invasive (arterial blood gas analysis - pH, PaO2, PaCO2, SaO2) measurements

Possible biases and confounding variables could be caused by hypothermia of participant, by sphygmomanometer cuff pressure on the same arm where blood samples are drawn and by prolonged time of arterial blood analysis. These difficulties can be bypassed by: adjustment of room temperature where analgo-sedation is performed, blood pressure measuring on opposite arm from where samples of blood are taken and by arterial blood gas analysis without delay.

Basic data analyses will be performed by statistician. Sample size is determined by statistic computing web program: http://www.stat.ubc.ca/~rollin/stats/ssize used statistic test Inference for Proportions: Comparing Two Independent Samples. Assessment of sample size is computed for two independent samples with assumption of clinically significant difference in patients' oxygenation: ≤11 and ≥14.4 kPa with delta 4.4. Statistical significance of difference will be inferred with 5% α-error, 50% β-error and study power 0.80. Calculated size of sample is: 21 participant pro subgroup (total of 126 participants).

Investigators expect no changes to methods after trial commencement. All potential unwanted events which may happen during analgo-sedation and colonoscopy that could cause deviation from this trial's protocol will be reason for exclusion of participant from this trial. If circumstances change, anesthesiologist responsible for application of anesthesia will carry out procedure in way which is in patients' best interest.

ELIGIBILITY:
Inclusion Criteria:

* normal weight ASA I patient
* normal weight ASA II patient
* normal weight ASA III patient
* intravenous analgo-sedation
* elective colonoscopy
* colorectal tumors.

Exclusion Criteria:

* obese patients
* emergency colonoscopy
* diseases of peripheral blood vessels
* hematological diseases
* psychiatric diseases
* sideropenic anemia
* patients' refusal
* ongoing chemotherapy or irradiation
* propofol allergies
* fentanyl allergies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of peripheral blood oxygenation (SpO2), | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Peripheral blood saturation (SpO2):
  Normal range ≥ 92% Acceptable deflection from normal values of peripheral blood saturation (SpO2) significant for hypoxemia is < 92%, while all values above will be considered normal.
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Change of arterial blood saturation (PaO2) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Partial pressure of oxygen (PaO2):
  Normal range: ≥11 kPa partial pressure of oxygen (PaO2), ≥ 11 kPa PaO2 will be considered normal, while all values below are considered significant for hypoxemia.
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.

SECONDARY OUTCOMES:
Change of partial pressure of CO2 (PaCO2) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Partial pressure of CO2 (PaCO2):
  Normal range: 4.7 - 6.4 kPa. Acceptable deflection from normal values significant for hypercapnia: PaCO2 ≥ 6 kPa
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Change of pH (pH) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  pH value of arterial blood sample :
  Normal values: 7.35 - 7.45. Acceptable deflection from normal values significant for acidosis: pH <7.35.
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Change of normopnea (FoB) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Frequency of breathing. (FoB/min - number of breaths per minute). Normal range: 12 - 20 breaths per minute. Bradypnoea will be noted when number of breaths is less than 12 breaths/min.
Change of frequency of desaturation (fDE) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Frequency of desaturation during time of analgo-sedation: (fDE/min, SpO2<92%). Normal range: fDE ≤1/30, up to one episode of desaturation from the start to the end of analgo-sedation. Acceptable deflection from normal range: more than one desaturation in 30 minutes.
Change of duration of desaturation (DE/min) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Duration of desaturation (DE/min). Normal range: up to one minute. Duration of desaturation longer then one minute will be considered as insufficient ventilation.
Change of frequency of bradypnoea during analgo-sedation (fBRP/min) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Frequency of bradypnoea during analgo-sedation (fBRP/min), Normal range: fBRP ≤1/30, up to one episode of bradypnoea from the start to the end of analgo-sedation. Acceptable deflection from normal range: > one episode of bradypnoea during 30 minutes.
Change of heart rate (HR/min) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Heart rate (HR/min): normal range 60 -100/min. Acceptable deflection from normal values is < 60 heartbeats/min significant for bradycardia, while all values up to 100 heartbeats per minute will be considered normal.
Change of mean arterial pressure (MAP) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Mean arterial pressure (MAP): normal range: 65 -110 mmHg Acceptable deflection from normal values is < 65 mmHg - significant for hypotension.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Behrens A, Ell C; Studiengruppe ALGK-ProSed. [Safety of sedation during gastroscopy and colonoscopy in low-risk patients - results of a retrospective subgroup analysis of a registry study including over 170 000 endoscopies]. Z Gastroenterol. 2016 Aug;54(8):733-9. doi: 10.1055/s-0042-108655. Epub 2016 Aug 16. German. PMID 27529524
- [Background] Anand GW, Heuss LT. Feasibility of breath monitoring in patients undergoing elective colonoscopy under propofol sedation: A single-center pilot study. World J Gastrointest Endosc. 2014 Mar 16;6(3):82-7. doi: 10.4253/wjge.v6.i3.82. PMID 24634712
- [Background] Becker DE, Haas DA. Management of complications during moderate and deep sedation: respiratory and cardiovascular considerations. Anesth Prog. 2007 Summer;54(2):59-68; quiz 69. doi: 10.2344/0003-3006(2007)54[59:MOCDMA]2.0.CO;2. PMID 17579505
- [Background] Frat JP, Goudet V, Girault C. [High flow, humidified-reheated oxygen therapy: a new oxygenation technique for adults]. Rev Mal Respir. 2013 Oct;30(8):627-43. doi: 10.1016/j.rmr.2013.04.016. Epub 2013 May 29. French. PMID 24182650
- [Background] Booth AWG, Vidhani K, Lee PK, Thomsett CM. SponTaneous Respiration using IntraVEnous anaesthesia and Hi-flow nasal oxygen (STRIVE Hi) maintains oxygenation and airway patency during management of the obstructed airway: an observational study. Br J Anaesth. 2017 Mar 1;118(3):444-451. doi: 10.1093/bja/aew468. PMID 28203745
- [Background] Schumann R, Natov NS, Rocuts-Martinez KA, Finkelman MD, Phan TV, Hegde SR, Knapp RM. High-flow nasal oxygen availability for sedation decreases the use of general anesthesia during endoscopic retrograde cholangiopancreatography and endoscopic ultrasound. World J Gastroenterol. 2016 Dec 21;22(47):10398-10405. doi: 10.3748/wjg.v22.i47.10398. PMID 28058020
- [Background] Nagata K, Morimoto T, Fujimoto D, Otoshi T, Nakagawa A, Otsuka K, Seo R, Atsumi T, Tomii K. Efficacy of High-Flow Nasal Cannula Therapy in Acute Hypoxemic Respiratory Failure: Decreased Use of Mechanical Ventilation. Respir Care. 2015 Oct;60(10):1390-6. doi: 10.4187/respcare.04026. Epub 2015 Jun 23. PMID 26106206
- [Background] Ni YN, Luo J, Yu H, Liu D, Ni Z, Cheng J, Liang BM, Liang ZA. Can High-flow Nasal Cannula Reduce the Rate of Endotracheal Intubation in Adult Patients With Acute Respiratory Failure Compared With Conventional Oxygen Therapy and Noninvasive Positive Pressure Ventilation?: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):764-775. doi: 10.1016/j.chest.2017.01.004. Epub 2017 Jan 13. PMID 28089816
- [Background] Morris K. Revising the Declaration of Helsinki. Lancet. 2013 Jun 1;381(9881):1889-90. doi: 10.1016/s0140-6736(13)60951-4. No abstract available. PMID 23734387
- [Background] Moher D, Schulz KF, Altman DG; CONSORT Group. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Clin Oral Investig. 2003 Mar;7(1):2-7. doi: 10.1007/s00784-002-0188-x. Epub 2003 Jan 31. PMID 12673431
- See also: American Society of Anesthesiologists (ASA). ASA physical status classification system 2014 Oct [internet]. Schaumburg, Illinois, USA: ASA;2014. — http://www.asahq.org/resources/clinical-information/asa-physical-status-classification-system
- See also: Programiz [internet].Kupandole, Nepal: Parewa Labs Pvt. Ltd. [cited 2018 Sept17]. Flowchart in programming. Available from: — http://www.programiz.com/article/flowchart-programming